CLINICAL TRIAL: NCT03947112
Title: Physical Activity Level of Norwegian Boys with Duchenne Muscular Dystrophy - a Cross Sectional Study
Brief Title: Physical Activity Level of Norwegian Boys with Duchenne Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Collaborators: Norwegian School of Sport Sciences (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/260
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2021-11

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Physical activity level
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Norwegian population with Duchenne Muscular Dystrophy (DMD): Boys with DMD.
  Interventions: Behavioral: Physical activity registration

INTERVENTIONS:
Behavioral: Physical activity registration — At start, participants and parents fills out a Self-report questionnaire and the UngKan-3 Questionnaire, before a seven day physical activity registration takes place by use og ActiGraph. A physical activity diary are filled out every evening while the physical activity registration takes places.
  Other Names: Self-report Questionnaire; Physical activity diary; UngKan-3 Questionnaire

SUMMARY:
The aim of this population based study is to examine, quantify and describe physical activity level in Norwegian boys with DMD, and to compare the level of physical activity level between boys with DMD and age matched healthy boys. A co-project will validate ActiGraph accelerometry to measure physical activity in boys with DMD.

DETAILED DESCRIPTION:
International guidelines recommend regular physical activity for boys with DMD, and participation in physical activity plays a key role in the management. Paradoxically, patients with severe neuromuscular disease like DMD, have considerable limitations to participate in such activities. Limitation may be muscle weakness, pain, fatigue, reduced mobility and overall function, and also limited knowledge of physical activity benefits among health care personnel. Limited participation leads to a sedentary lifestyle, and gradual under-use of still functioning muscles may cause secondary deterioration in DMD.

The current physical activity level amongst Norwegian DMD's are unknown, and physical activity registration and self-reported questionnaire will be examined in this study.

ELIGIBILITY:
Inclusion Criteria:

* Boys with conclusive diagnosis of Duchenne Muscular disease, attending Norwegian pediatric rehabilitation clinics.
* Signed written consent
* Able to answer questionnaires with help from parents, care giver(s) or health care professional with regular follow up of the participants.

Exclusion Criteria:

* Lack of consent.
* Language difficulties
* Cognitive dysfunction or mental retardation leading to difficulties in answering the questionnaires adequately

Ages: 6 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — DMD is X-linked disease
Study Population: Study population will be requited from all the Norwegian regional pediatric rehabilitation centre's out patient clinics. Verbal and written information about the study will be provided if inclution criteria to be met.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Physical activity registration | Seven days
  An Actigraph will be provided and worn at pre set time frame (Seven days including weekend). Data extracted are counts per minutes, and are measurements of movement performed in both vertical and horizontal axis. The counts will be used to quantify the time the participant is inactive, low, moderate and / or in vigorous physical active.

SECONDARY OUTCOMES:
Leisure time physical activity | Day 1
  The UngKan-3 questionnaire is a self-reported/parent-reported instrument, developed to measure leisure time physical activity, diet, media habits and sleep routine. The questionnaire is former used in a national cross-sectional survey amongst Norwegian school students, developed by the Norwegian School of Sport Sciences and Norwegian Institute of Public Health.
Self-Reported Questionnaire | Day 1
  Self-administrated questionnaire developed to describe participants function, on-going treatment, movement aid, types of physical activities

OTHER OUTCOMES:
Physical Activity diary | Day 1
  During physical activity registration with use of ActiGraph monitor, the participants and parents are asked to fill out a diary, describing type of physical activity been performed, for how long the physical activity was performed, how tired the participants became, and how did the participant enjoy the activity being performed. In addition the participants is asked to give a summary of the week regarding to name the most enjoyable activity this week and the reason why, and to describe if there occurred something unusual that increased or decreased their physical activity level more than regular.

CONTACTS AND LOCATIONS:
Overall Officials: Tiina M Andersen, PhD, Principal Investigator — Department of Physiotherapy, Haukeland University Hospital, Bergen, Norway
Locations (1):
- Haukeland University Hospital, Bergen, Hordaland, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heutinck L, Kampen NV, Jansen M, Groot IJ. Physical Activity in Boys With Duchenne Muscular Dystrophy Is Lower and Less Demanding Compared to Healthy Boys. J Child Neurol. 2017 Apr;32(5):450-457. doi: 10.1177/0883073816685506. Epub 2017 Jan 23. PMID 28112012
- [Background] Birnkrant DJ, Bushby K, Bann CM, Apkon SD, Blackwell A, Brumbaugh D, Case LE, Clemens PR, Hadjiyannakis S, Pandya S, Street N, Tomezsko J, Wagner KR, Ward LM, Weber DR; DMD Care Considerations Working Group. Diagnosis and management of Duchenne muscular dystrophy, part 1: diagnosis, and neuromuscular, rehabilitation, endocrine, and gastrointestinal and nutritional management. Lancet Neurol. 2018 Mar;17(3):251-267. doi: 10.1016/S1474-4422(18)30024-3. Epub 2018 Feb 3. PMID 29395989